CLINICAL TRIAL: NCT00229957
Title: Rehabilitation in Primary Care: A Project to Maximize the Health Status of Adults With Chronic Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 04-052; G03-02572
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Results first posted 2010-07-07 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2009-09

CONDITIONS: Chronic Disease; Hypertension; Back Pain; Obesity; Arthritis
Keywords: Occupational therapy; Physical therapy techniques; Primary health care; Chronic disease; Rehabilitation; Disease management; Self care
MeSH Terms: conditions — Chronic Disease; Hypertension; Back Pain; Obesity; Arthritis | interventions — Occupational Therapy; Physical Therapy Modalities; Self-Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Intervention
  Interventions: Behavioral: Occupational therapy; Behavioral: Physiotherapy; Behavioral: Self-management
- Control (No Intervention): Control group received usual care in primary care.

INTERVENTIONS:
Behavioral: Occupational therapy
  Arms: Intervention
Behavioral: Physiotherapy
  Arms: Intervention
Behavioral: Self-management
  Arms: Intervention

SUMMARY:
The purpose of the study is to determine whether occupational therapy and physiotherapy delivered in a primary care setting to adults with chronic illness is effective in improving health.

DETAILED DESCRIPTION:
Primary health care is changing so that people receive the care that they need at the front line. Rehabilitation has been identified as one service that should be offered in primary care, to address the needs of adults who have or are at risk of poor health from chronic conditions such as arthritis, heart disease and depression.

Two full time therapists (one physiotherapist and one occupational therapist) will offer rehabilitation to a sample of 170 adults with chronic illness over an 18 month period (170 people will also be enrolled in a control group) at the Stonechurch Family Health Centre. Key outcomes include health, hospital admissions and emergency room visits.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 chronic condition
* 3 visits to family physician in the past year

Exclusion Criteria:

* None

Min Age: 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2004-06; Primary Completion 2006-08 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Letts, PhD, Principal Investigator — McMaster University; Julie Richardson, PhD, Principal Investigator — McMaster University
Locations (1):
- Stonechurch Family Health Centre, 549 Stonechurch Rd. E., Hamilton, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants recruited from a family health practice.
Groups:
- Intervention Group: A rehabilitation multi-component intervention delivered by a physiotherapist and occupational therapist in a primary care setting included collaborative goal setting for rehabilitation needs, a six-week chronic disease self-management workshop, referral to community programs and a web-based education programme.
- Control Group: Usual care from the primary health care team which did not include physiotherapy or occupational therapy.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 152 | 151
Completed | 132 | 139
Not Completed | 20 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 152 | 151 | 303
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 86 | 86 | 172
  >=65 years | 66 | 65 | 131
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 94 | 192
  Male | 54 | 57 | 111

OUTCOME MEASURES:

1. Primary Outcome: SF-36 Physical Component
Description: health related quality of life. Minimum: 0; Maximum 100.
Time Frame: 15 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 132 | 139
units on a scale | 42.6 (11.8) | 43.1 (11.9)

2. Secondary Outcome: Use of Hospital Services
Description: self report use of hospital service
Time Frame: baseline, 15 months
Reporting Status: Not Posted, anticipated posting 2009-07
Measure: Mean (Standard Deviation); unit: planned hospital days, ER visits

3. Secondary Outcome: Independence in Activities of Daily Living (ADLs) and Instrumental Activities of Daily Living (IADLs)
Description: Late Life Function and Disability Instrument: A measure of disability and functional limitations in older adults. (Score range 0-100 with 100 representing better ability and less disability/functional limitation)
Time Frame: baseline, 15 months
Reporting Status: Not Posted, anticipated posting 2009-08
Measure: Mean (Standard Deviation); unit: units on a scale

4. Secondary Outcome: Functional Limitations
Description: Late Life Function and Disability Instrument: A measure of functional limitations and disability in older adults.
Time Frame: baseline, 15 months
Reporting Status: Not Posted, anticipated posting 2009-08
Measure: Mean (Standard Deviation); unit: units on a scale

5. Secondary Outcome: Falls and Injuries
Description: self-reported number of falls in last 6 months
Time Frame: baseline, 15 months
Reporting Status: Not Posted, anticipated posting 2009-08
Measure: Mean; unit: number of falls

6. Secondary Outcome: HOME Falls and Accident Screening Tool (FAST)
Description: This is a home assessment of safety hazards for falls present in the individual's home. This tool helps to identify seniors at risk of falls. Score 0-25.
Time Frame: baseline, 15 months
Reporting Status: Not Posted, anticipated posting 2009-08
Measure: Mean (Standard Deviation); unit: number

7. Secondary Outcome: Self-management and Self-efficacy
Description: Individual's self-reported ability to carry out behaviours to self-manage their health condition, and their confidence level in being able to carry out these behaviours. (Score range 0= not confident at all, 10= totally confident).
Time Frame: baseline, 15 months
Reporting Status: Not Posted, anticipated posting 2009-08
Measure: Mean (Standard Deviation); unit: units on a scale

8. Secondary Outcome: Physical Abilities (Strength, Balance)
Description: Grip strength was measured using a JAMAR hand grip dynamometer (in kilograms). The Lower Extremity Function test is a battery of three tests used to measure lower extremity function and balance: a balance test, 8 foot walk test, and repetitive standing from a chair. A performance summary score is created by adding the number of seconds achieved on the balance test, the number of seconds to walk 8 feet and the number of seconds it takes the person to stand up from a chair five times consecutively (no maximum score exists on this measure).
Time Frame: baseline, 15 months
Reporting Status: Not Posted, anticipated posting 2009-08
Measure: Mean (Standard Deviation); unit: kilograms, seconds

9. Secondary Outcome: Patient Satisfaction Questionnaire - 18 (Modified)
Description: Patient satisfaction with the care they received. (Score range 0-5)
Time Frame: 15 months
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: units on a scale

ADVERSE EVENTS:
Arm/Group | Intervention Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/152 | 0/151
Other Adverse Events (participants affected / at risk) | 0/152 | 0/151

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No